CLINICAL TRIAL: NCT00945230
Title: Analysis of Post Surgical Response in A Fifty-Six Year Old Female With An Incidental Large Left Anterior Cranial Fossa Meningioma
Brief Title: Actigraphic Measurement of a Neurosurgical Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Psychopharmacology Institute (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Bill J. Duke, M.A., Ph.D., ABMPP, Child Psychopharmacology Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Act2NS
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Sleep Disorders; Circadian Rhythm; Pain; Rehabilitation; Mood Lability
Keywords: Neurosurgical outcome; Actigraphy; Treatment Response Measurement
MeSH Terms: conditions — Sleep Wake Disorders; Pain | interventions — Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Actigraphic Neurosurgical Outcomes (Experimental): Actigraphic measurements that will be obtained by attaching the actigraphic watch device to the individual's non-dominant wrist and operationally defined repeated observational measurements. All measurements will continue through a baseline period and continue through the identified post surgical period. Actigraphic measurements will occur every 30 seconds with brief periods of non-measurement during the actual neurosurgical procedure and periods when the actigraphic device has reached storage capacity (approximately every 22 days) when data is retrieved and the device prepared resume measurements.
  Interventions: Procedure: Re-section of a large left anterior cranial fossa meningioma

INTERVENTIONS:
Procedure: Re-section of a large left anterior cranial fossa meningioma — Neurosurgical re-section of an incidental large left anterior cranial fossa meningioma
  Other Names: Actigraphy

SUMMARY:
The study examines and illustrates the utility of utilizing actigraphic measurements to assess treatment response.

DETAILED DESCRIPTION:
Actigraphic measurements, repeated verbal fluency and multi-symptom operationally defined observations will be recorded for an 11 to 12 day baseline period and continued following neurosurgical tumor resection until a repeat MRI is completed three months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of incidental meningioma
* Single subject preparing to receive neurosurgical intervention

Exclusion Criteria:

* Inability to wear actigraphy device

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pre and Post Actigraphic and Systematic Observation Scale measurements | March 15, 2009-June 20, 2009

CONTACTS AND LOCATIONS:
Overall Officials: Bill J Duke, M.A., Ph.D., Principal Investigator — Child Psychopharmacology Institute
Locations (1):
- Child Psychopharmacology Institute, Fargo, North Dakota, United States